CLINICAL TRIAL: NCT05366491
Title: Serum Human IL-38 Levels in Asthmatic Children
Brief Title: IL-38 Evaluation as a Biomarker in Pediatric Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Kamal, Assistant professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MS-25-2020
Record Dates: First submitted 2022-05-05; First posted 2022-05-09 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bronchial asthma patients (Active Comparator): patients diagnosed with bronchial asthma
  Interventions: Diagnostic Test: Il-38 serum level
- healthy controls (Active Comparator): healthy subjects with age and sex matched to bronchial asthma patients
  Interventions: Diagnostic Test: Il-38 serum level

INTERVENTIONS:
Diagnostic Test: Il-38 serum level — measurement of serum levels of IL-38

SUMMARY:
The aim of this study is to investigate the associations between serum IL-38 levels and different variables of asthma in children such as laboratory variables, pulmonary function test results, the diagnosis of asthma, and in correlation with disease severity.

ELIGIBILITY:
Inclusion Criteria:

* patients fulfilled the criteria of the Global Initiative for Asthma (GINA)
* Age group:6-14 years

Exclusion Criteria:

* Malignancy
* Chronic inflammatory diseases

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
serum IL-38 levels | within 6 months
  Measurement of Interleukin 38 in sera of all study subjects by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Kamal, Ass prof, Principal Investigator — Assistant professor
Locations (1):
- Asmaa Kamal, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No